CLINICAL TRIAL: NCT03425487
Title: Mindfulness-based and Compassion-based Interventions in Anxious-Depressive Symptomatology in Mental Health Services: A Randomized Controlled Trial
Brief Title: Mindfulness-based and Compassion-based Interventions in Anxious-Depressive Symptomatology in Mental Health Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Miguel Servet (Other)
Responsible Party: Principal Investigator, Javier Garcia Campayo, Principal Investigator, Hospital Miguel Servet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7/2017
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Anxious-Depressive
Keywords: Mindfulness; Compassion; Mental Health Services

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MBSR+TAU (Experimental): Mindfulness based Intervention (MBSR) + Usual specialized treatment in mental health. MBSR consists of 8 weekly groupal sessions of 150 minutes/session (10-16 people). Written material and sound recordings will be offered as support elements. The estimated duration of the program is two months.
  Interventions: Behavioral: Mindfulness based Intervention
- ABCT+TAU (Experimental): Compassion based Intervention (ABCT) + Usual specialized treatment in mental health. ABCT consists of 8 weekly groupal sessions of 120 minutes/session (10-16 people). Written material and sound recordings will be offered as support elements. The estimated duration of the program is two months.
  Interventions: Behavioral: Compassion based Intervention
- TAU (Active Comparator): Usual specialized treatment in mental health (psychological or/and psychiatric)
  Interventions: Other: TAU

INTERVENTIONS:
Behavioral: Mindfulness based Intervention — MBSR consists of 8 weekly groupal sessions of 150 minutes/session (10-16 people). Written material and sound recordings will be offered as support elements. The estimated duration of the program is two months
  Arms: MBSR+TAU
Behavioral: Compassion based Intervention — ABCT consists of 8 weekly groupal sessions of 120 minutes/session (10-16 people). Written material and sound recordings will be offered as support elements. The estimated duration of the program is two months.
  Arms: ABCT+TAU
Other: TAU — Usual specialized treatment in mental health (psychological or/and psychiatric)
  Arms: TAU

SUMMARY:
The aim of this study is to assess and compare the benefits of twopsychological interventions added to the usual treatment of patients whocome to mental health. Patients will be randomly assigned to the followingconditions: Mindfulness-Based Stress Reduction (MBSR), Attachment-BasedCompassion Therapy (ABCT) and a Treatment As Usual (TAU) Group. Theparticipants in the two psychological intervention groups will also receive usualpsychological/psychiatric treatment managed by their specialist. Mindfulnessand Compassion groups will be composed of 33 participants each, and TAU group will be composed of 64 participants (total sample n = 130).

The principal hypothesis is that 'ABCT + TAU' will be more effective than'MBSR + TAU' for treating depressive and/or anxiety symptoms in patients attending mental health settings. Secondary hypothesis are: 1) 'MBSR + TAU'and 'ABCT + TAU' will be more effective than 'TAU alone' for treatinganxiety and/or depressive symptoms in patients attending mental health settings; 2) mindfulness will be a mediator of the 'MBSR + TAU' program improvements, while self-compassion will be a mediator of the corresponding'ABCT + TAU'; and 3) 'ABCT + TAU' will present more cost-effectiveness than 'MBSR + TAU' and both ABCT + TAU' and 'MBSR + TAU' programs will present more cost-effectiveness than TAU alone.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old.
* Depressive and/or anxious disorder, or adjustment disorder with depressive or/and anxious symptomatology, according to clinical criteria based on Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
* Disorder of mild or moderate severity according to clinical criteria (based on DSM-5).
* Understand perfectly spoken and written Spanish.
* Grant a written informed consent form

Exclusion Criteria:

* To have done any type of meditative/contemplative practice during the previous year.
* Any diagnose of disease that may affect central nervous system (brain pathology, traumatic brain injury, dementia, etc.).
* Other psychiatric diagnoses or acute psychiatric illness (substance dependence or abuse, history of schizophrenia or other psychotic disorders, eating disorders, etc.).
* Any medical, infectious or degenerative disease that may affect mood.
* Presence of delusional ideas or hallucinations consistent or not with mood, and suicide risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scales | Baseline
  In the MBSR based intervention group. This scale is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The range for each subescale is 0-21 (But this scores will need to be multiplied by 2 to calculate the final score). This questionnaire also gives us a one-dimensional global measure of emotional distress that will be considered as the main study outcome. It is composed by all the 21 items configuring a general factor, and it will be taken as a continuous dimensional variable that ranges from 0 to 126.
Depression Anxiety Stress Scales | Baseline
  In the ABCT based intervention group. This scale is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The range for each subescale is 0-21 (But this scores will need to be multiplied by 2 to calculate the final score). This questionnaire also gives us a one-dimensional global measure of emotional distress that will be considered as the main study outcome. It is composed by all the 21 items configuring a general factor, and it will be taken as a continuous dimensional variable that ranges from 0 to 126.
Depression Anxiety Stress Scales | Baseline
  In the TAU control group. This scale is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The range for each subescale is 0-21 (But this scores will need to be multiplied by 2 to calculate the final score). This questionnaire also gives us a one-dimensional global measure of emotional distress that will be considered as the main study outcome. It is composed by all the 21 items configuring a general factor, and it will be taken as a continuous dimensional variable that ranges from 0 to 126.
Depression Anxiety Stress Scales | Post-treatment 8 weeks from baseline in 8 weeks MBSR intervention group
  In the MBSR based intervention group. This scale is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The range for each subescale is 0-21 (But this scores will need to be multiplied by 2 to calculate the final score). This questionnaire also gives us a one-dimensional global measure of emotional distress that will be considered as the main study outcome. It is composed by all the 21 items configuring a general factor, and it will be taken as a continuous dimensional variable that ranges from 0 to 126.
Depression Anxiety Stress Scales | Post-treatment 8 weeks from baseline in 8 weeks ABCT intervention group
  In the ABCT based intervention group. This scale is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The range for each subescale is 0-21 (But this scores will need to be multiplied by 2 to calculate the final score). This questionnaire also gives us a one-dimensional global measure of emotional distress that will be considered as the main study outcome. It is composed by all the 21 items configuring a general factor, and it will be taken as a continuous dimensional variable that ranges from 0 to 126.
Depression Anxiety Stress Scales | Post-treatment 8 weeks from baseline in TAU control group
  In the TAU control group. This scale is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The range for each subescale is 0-21 (But this scores will need to be multiplied by 2 to calculate the final score). This questionnaire also gives us a one-dimensional global measure of emotional distress that will be considered as the main study outcome. It is composed by all the 21 items configuring a general factor, and it will be taken as a continuous dimensional variable that ranges from 0 to 126.
Depression Anxiety Stress Scales | Six-months follow-up
  In the MBSR based intervention group. This scale is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The range for each subescale is 0-21 (But this scores will need to be multiplied by 2 to calculate the final score). This questionnaire also gives us a one-dimensional global measure of emotional distress that will be considered as the main study outcome. It is composed by all the 21 items configuring a general factor, and it will be taken as a continuous dimensional variable that ranges from 0 to 126.
Depression Anxiety Stress Scales | Six-months follow-up
  In the ABCT based intervention group. This scale is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The range for each subescale is 0-21 (But this scores will need to be multiplied by 2 to calculate the final score). This questionnaire also gives us a one-dimensional global measure of emotional distress that will be considered as the main study outcome. It is composed by all the 21 items configuring a general factor, and it will be taken as a continuous dimensional variable that ranges from 0 to 126.
Depression Anxiety Stress Scales | Six-months follow-up
  In the TAU control group. This scale is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The range for each subescale is 0-21 (But this scores will need to be multiplied by 2 to calculate the final score). This questionnaire also gives us a one-dimensional global measure of emotional distress that will be considered as the main study outcome. It is composed by all the 21 items configuring a general factor, and it will be taken as a continuous dimensional variable that ranges from 0 to 126.

SECONDARY OUTCOMES:
Sociodemographic data such as gender, age, marital status, education, occupation, economical level | Baseline
  In the MBSR based intervention group
Sociodemographic data such as gender, age, marital status, education, occupation, economical level | Baseline
  In the ABCT based intervention group
Sociodemographic data such as gender, age, marital status, education, occupation, economical level | Baseline
  In the TAU control group
Five Facet Mindfulness Questionnaire | Baseline
  In the MBSR based intervention group. The FFMQ is a 39-item questionnaire that measures five facets of mindfulness: observe (8 items), describe (8 items), actaware (8 items), nonjudge (8 items) and nonreact (7 items). The range score for each subescale is: "observe" (40 points); "describe" (40 points); "actaware" (40 points); "nonjudge"(40 points); "nonreact" (35 points). For all subscales, a high score is considered to be more presence of the construct. Finally, the subscales can be summed to obtain a general score.
Five Facet Mindfulness Questionnaire | Baseline
  In the ABCT based intervention group. The FFMQ is a 39-item questionnaire that measures five facets of mindfulness: observe (8 items), describe (8 items), actaware (8 items), nonjudge (8 items) and nonreact (7 items). The range score for each subescale is: "observe" (40 points); "describe" (40 points); "actaware" (40 points); "nonjudge"(40 points); "nonreact" (35 points). For all subscales, a high score is considered to be more presence of the construct. Finally, the subscales can be summed to obtain a general score.
Five Facet Mindfulness Questionnaire | Baseline
  In the TAU control group. The FFMQ is a 39-item questionnaire that measures five facets of mindfulness: observe (8 items), describe (8 items), actaware (8 items), nonjudge (8 items) and nonreact (7 items). The range score for each subescale is: "observe" (40 points); "describe" (40 points); "actaware" (40 points); "nonjudge"(40 points); "nonreact" (35 points). For all subscales, a high score is considered to be more presence of the construct. Finally, the subscales can be summed to obtain a general score.
Five Facet Mindfulness Questionnaire | Post-treatment 8 weeks from baseline in 8 weeks MBSR intervention group
  In the MBSR based intervention group. The FFMQ is a 39-item questionnaire that measures five facets of mindfulness: observe (8 items), describe (8 items), actaware (8 items), nonjudge (8 items) and nonreact (7 items). The range score for each subescale is: "observe" (40 points); "describe" (40 points); "actaware" (40 points); "nonjudge"(40 points); "nonreact" (35 points). For all subscales, a high score is considered to be more presence of the construct. Finally, the subscales can be summed to obtain a general score.
Five Facet Mindfulness Questionnaire | Post-treatment 8 weeks from baseline in 8 weeks ABCT intervention group
  In the ABCT based intervention group. The FFMQ is a 39-item questionnaire that measures five facets of mindfulness: observe (8 items), describe (8 items), actaware (8 items), nonjudge (8 items) and nonreact (7 items). The range score for each subescale is: "observe" (40 points); "describe" (40 points); "actaware" (40 points); "nonjudge"(40 points); "nonreact" (35 points). For all subscales, a high score is considered to be more presence of the construct. Finally, the subscales can be summed to obtain a general score.
Five Facet Mindfulness Questionnaire | Post-treatment 8 weeks from baseline in TAU control group
  In the TAU group control. The FFMQ is a 39-item questionnaire that measures five facets of mindfulness: observe (8 items), describe (8 items), actaware (8 items), nonjudge (8 items) and nonreact (7 items). The range score for each subescale is: "observe" (40 points); "describe" (40 points); "actaware" (40 points); "nonjudge"(40 points); "nonreact" (35 points). For all subscales, a high score is considered to be more presence of the construct. Finally, the subscales can be summed to obtain a general score.
Five Facet Mindfulness Questionnaire | Six-months follow-up
  In the MBSR based intervention group. The FFMQ is a 39-item questionnaire that measures five facets of mindfulness: observe (8 items), describe (8 items), actaware (8 items), nonjudge (8 items) and nonreact (7 items). The range score for each subescale is: "observe" (40 points); "describe" (40 points); "actaware" (40 points); "nonjudge"(40 points); "nonreact" (35 points). For all subscales, a high score is considered to be more presence of the construct. Finally, the subscales can be summed to obtain a general score.
Five Facet Mindfulness Questionnaire | Six-months follow-up
  In the ABCT based intervention group. The FFMQ is a 39-item questionnaire that measures five facets of mindfulness: observe (8 items), describe (8 items), actaware (8 items), nonjudge (8 items) and nonreact (7 items). The range score for each subescale is: "observe" (40 points); "describe" (40 points); "actaware" (40 points); "nonjudge"(40 points); "nonreact" (35 points). For all subscales, a high score is considered to be more presence of the construct. Finally, the subscales can be summed to obtain a general score.
Five Facet Mindfulness Questionnaire | Six-months follow-up
  In the TAU group control. The FFMQ is a 39-item questionnaire that measures five facets of mindfulness: observe (8 items), describe (8 items), actaware (8 items), nonjudge (8 items) and nonreact (7 items). The range score for each subescale is: "observe" (40 points); "describe" (40 points); "actaware" (40 points); "nonjudge"(40 points); "nonreact" (35 points). For all subscales, a high score is considered to be more presence of the construct. Finally, the subscales can be summed to obtain a general score.
Self-Compassion Scale | Baseline
  In the MBSR based intervention group. This scale is currently the only self-report instrument to measure self-compassion. The SCS is divided into six subscales: 4-item Self-Kindness; 4-item Self-Judgment; 4-item Common Humanity; 4-item Isolation; 4-item Mindfulness; and 4-item Over-Identification. The items can be rated on a five-point likert scale with 1 indicating almost never and 5 indicating almost always. After reversing the negatively formulated items, a total score can be calculated, which may range from 24 to 120, with higher scores indicating greater self-compassion.
Self-Compassion Scale | Baseline
  In the ABCT based intervention group. This scale is currently the only self-report instrument to measure self-compassion. The SCS is divided into six subscales: 4-item Self-Kindness; 4-item Self-Judgment; 4-item Common Humanity; 4-item Isolation; 4-item Mindfulness; and 4-item Over-Identification. The items can be rated on a five-point likert scale with 1 indicating almost never and 5 indicating almost always. After reversing the negatively formulated items, a total score can be calculated, which may range from 24 to 120, with higher scores indicating greater self-compassion.
Self-Compassion Scale | Baseline
  In the TAU group control. This scale is currently the only self-report instrument to measure self-compassion. The SCS is divided into six subscales: 4-item Self-Kindness; 4-item Self-Judgment; 4-item Common Humanity; 4-item Isolation; 4-item Mindfulness; and 4-item Over-Identification. The items can be rated on a five-point likert scale with 1 indicating almost never and 5 indicating almost always. After reversing the negatively formulated items, a total score can be calculated, which may range from 24 to 120, with higher scores indicating greater self-compassion.
Self-Compassion Scale | Post-treatment 8 weeks from baseline in 8 weeks MBSR intervention group
  In the MBSR based intervention group. This scale is currently the only self-report instrument to measure self-compassion. The SCS is divided into six subscales: 4-item Self-Kindness; 4-item Self-Judgment; 4-item Common Humanity; 4-item Isolation; 4-item Mindfulness; and 4-item Over-Identification. The items can be rated on a five-point likert scale with 1 indicating almost never and 5 indicating almost always. After reversing the negatively formulated items, a total score can be calculated, which may range from 24 to 120, with higher scores indicating greater self-compassion.
Self-Compassion Scale | Post-treatment 8 weeks from baseline in 8 weeks ABCT intervention group
  In the ABCT based intervention group. This scale is currently the only self-report instrument to measure self-compassion. The SCS is divided into six subscales: 4-item Self-Kindness; 4-item Self-Judgment; 4-item Common Humanity; 4-item Isolation; 4-item Mindfulness; and 4-item Over-Identification. The items can be rated on a five-point likert scale with 1 indicating almost never and 5 indicating almost always. After reversing the negatively formulated items, a total score can be calculated, which may range from 24 to 120, with higher scores indicating greater self-compassion.
Self-Compassion Scale | Post-treatment 8 weeks from baseline in TAU control group
  In the TAU group control. This scale is currently the only self-report instrument to measure self-compassion. The SCS is divided into six subscales: 4-item Self-Kindness; 4-item Self-Judgment; 4-item Common Humanity; 4-item Isolation; 4-item Mindfulness; and 4-item Over-Identification. The items can be rated on a five-point likert scale with 1 indicating almost never and 5 indicating almost always. After reversing the negatively formulated items, a total score can be calculated, which may range from 24 to 120, with higher scores indicating greater self-compassion.
Self-Compassion Scale | Six-months follow-up
  In the MBSR based intervention group. This scale is currently the only self-report instrument to measure self-compassion. The SCS is divided into six subscales: 4-item Self-Kindness; 4-item Self-Judgment; 4-item Common Humanity; 4-item Isolation; 4-item Mindfulness; and 4-item Over-Identification. The items can be rated on a five-point likert scale with 1 indicating almost never and 5 indicating almost always. After reversing the negatively formulated items, a total score can be calculated, which may range from 24 to 120, with higher scores indicating greater self-compassion.
Self-Compassion Scale | Six-months follow-up
  In the ABCT based intervention group. This scale is currently the only self-report instrument to measure self-compassion. The SCS is divided into six subscales: 4-item Self-Kindness; 4-item Self-Judgment; 4-item Common Humanity; 4-item Isolation; 4-item Mindfulness; and 4-item Over-Identification. The items can be rated on a five-point likert scale with 1 indicating almost never and 5 indicating almost always. After reversing the negatively formulated items, a total score can be calculated, which may range from 24 to 120, with higher scores indicating greater self-compassion.
Self-Compassion Scale | Six-months follow-up
  In the TAU group control. This scale is currently the only self-report instrument to measure self-compassion. The SCS is divided into six subscales: 4-item Self-Kindness; 4-item Self-Judgment; 4-item Common Humanity; 4-item Isolation; 4-item Mindfulness; and 4-item Over-Identification. The items can be rated on a five-point likert scale with 1 indicating almost never and 5 indicating almost always. After reversing the negatively formulated items, a total score can be calculated, which may range from 24 to 120, with higher scores indicating greater self-compassion.
EuroQol-5D. Health related quality of life | Baseline
  In the MBSR based intervention group. The EuroQol-5D is a standardized instrument for measuring generic health status. The construct "health status" is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using three-level scale.
EuroQol-5D. Health related quality of life | Baseline
  In the ABCT based intervention group. The EuroQol-5D is a standardized instrument for measuring generic health status. The construct "health status" is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using three-level scale.
EuroQol-5D. Health related quality of life | Baseline
  In the TAU group control. The EuroQol-5D is a standardized instrument for measuring generic health status. The construct "health status" is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using three-level scale.
EuroQol-5D. Health related quality of life | Post-treatment 8 weeks from baseline in 8 weeks MBSR intervention group
  In the MBSR based intervention group. The EuroQol-5D is a standardized instrument for measuring generic health status. The construct "health status" is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using three-level scale.
EuroQol-5D. Health related quality of life | Post-treatment 8 weeks from baseline in 8 weeks ABCT intervention group
  In the ABCT based intervention group. The EuroQol-5D is a standardized instrument for measuring generic health status. The construct "health status" is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using three-level scale.
EuroQol-5D. Health related quality of life | Post-treatment 8 weeks from baseline in TAU control group
  In the TAU group control. The EuroQol-5D is a standardized instrument for measuring generic health status. The construct "health status" is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using three-level scale.
EuroQol-5D. Health related quality of life | Six-months follow-up
  In the MBSR based intervention group. The EuroQol-5D is a standardized instrument for measuring generic health status. The construct "health status" is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using three-level scale.
EuroQol-5D. Health related quality of life | Six-months follow-up
  In the ABCT based intervention group. The EuroQol-5D is a standardized instrument for measuring generic health status. The construct "health status" is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using three-level scale.
EuroQol-5D. Health related quality of life | Six-months follow-up
  In the TAU group control. The EuroQol-5D is a standardized instrument for measuring generic health status. The construct "health status" is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using three-level scale.
Client Service Receipt Inventory (CSRI) | Baseline
  In the MBSR based intervention group
Client Service Receipt Inventory (CSRI) | Baseline
  In the ABCT based intervention group
Client Service Receipt Inventory (CSRI) | Baseline
  In the TAU group control
Client Service Receipt Inventory (CSRI) | Six-months follow-up
  In the MBSR based intervention group
Client Service Receipt Inventory (CSRI) | Six-months follow-up
  In the ABCT based intervention group
Client Service Receipt Inventory (CSRI) | Six-months follow-up
  In the TAU group control

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de la Plana, Castellon, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data generated by this trial will be made available upon reasonable request to researchers i) who provide a methodologically sound proposal and ii) whose proposed use of the data has been approved by an independent ethical review committee. The data sharing plan will include all of the individual anonymized and completely de-identified participant data collected during the trial, as well as other related documents such as the study protocol, the statistical analysis plan and the data dictionary with descriptive labels.
  The database will be encrypted and password protected.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available immediately following each publication with no end date and for any analytical purpose that is related to achieve aims in the original approved proposal.
Access Criteria: Passwords will be provided by the corresponding author to interested researchers that meet the both previously described criteria.

REFERENCES:
- [Derived] Collado-Navarro C, Navarro-Gil M, Perez-Aranda A, Lopez-Del-Hoyo Y, Garcia-Campayo J, Montero-Marin J. Effectiveness of mindfulness-based stress reduction and attachment-based compassion therapy for the treatment of depressive, anxious, and adjustment disorders in mental health settings: A randomized controlled trial. Depress Anxiety. 2021 Nov;38(11):1138-1151. doi: 10.1002/da.23198. Epub 2021 Jul 20. PMID 34288280
- [Derived] Montero-Marin J, Collado-Navarro C, Navarro-Gil M, Lopez-Montoyo A, Demarzo M, Herrera-Mercadal P, Barcelo-Soler A, Garcia-Campayo J. Attachment-based compassion therapy and adapted mindfulness-based stress reduction for the treatment of depressive, anxious and adjustment disorders in mental health settings: a randomised controlled clinical trial protocol. BMJ Open. 2019 Oct 8;9(10):e029909. doi: 10.1136/bmjopen-2019-029909. PMID 31597650